CLINICAL TRIAL: NCT04060186
Title: Balloninflation After Evacuation of Chronical Subdural Haematoma for Reduction of Hematoma Recurrrence: Randomized Controlled Study
Brief Title: Postoperative Balloninflation After Evacuation of cSDH
Acronym: BANISH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Marina Heibel, Study Nurse, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BANISH
Record Dates: First submitted 2019-08-06; First posted 2019-08-19 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Chronic Subdural Hematoma
Keywords: Recurrence rate of cSDH; Outcome
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloninflation Group (Active Comparator): Patient who will perform a balloninflation after operation
  Interventions: Procedure: Balloninflation
- Conservative Group (Sham Comparator): Patient without performing a balloninflation
  Interventions: Procedure: Balloninflation

INTERVENTIONS:
Procedure: Balloninflation — Patient will inflate into a ballon made by a handglove 2-3times/h from 8:00-20:00 after evacuation of chronic subdural hematoma.

SUMMARY:
In this prospective, randomized, multicenter trial shall patients with chronic subdural hematoma (cSDH) recruited, who were surgically treated. Initially, we would divide the patients randomized into two groups: Patients with supervised blow-maneuver and without. After surgical treatment of cSDH with insertion of a subdural drain, one group would perform a supervised blow maneuver ("Valsalva maneuver") every hour for five minutes from 10:00 to 20:00. In the other group, the standard care would be performed. The subdural drain would be explanted 2days after operation and a postoperative CT scan would routinely be performed. After hospital discharge, the patient would be rechecked in an ambulant setting and would receive CT scan as clinical standard. Recurrence of hematoma is defined as recurrent hematoma which should be reoperated. After 3 and 6 months we would evaluate the outcome of patients.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* surgically treated cSDH
* patients with an operatively implanted subdural drainage

Exclusion Criteria:

* age under 18 years
* Admission in critical clinical state, e.g. already to light unresponsive pupils for about 2 hours
* conservative treatment of cSDH
* patients without an operatively implanted subdural drainage
* patient cannot be consented
* participation in other clinical trials

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Recurrence Rate | 3 Months
  Reoperation of chronic subdural hematoma

SECONDARY OUTCOMES:
Neurological Functional Outcome | 6 Months
  Modified Rankin Scale (0-6) 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead. mRS0-3: favorable Outcome mRS: 4-6: unfavorable Outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Niederrad, Hesse, Germany